CLINICAL TRIAL: NCT04539067
Title: Effect of Controlled Ovarian Stimulation With H FSH and HHMg Vs HMG Alone on Oocyte and Embryo Quality in IcsI Patients
Brief Title: Effect of Controlled Ovarian Stimulation in Quality of Oocyte and Embryo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Marwa Bahgat Tarahony, Eygpt Minia, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 635_5/2020
Record Dates: First submitted 2020-08-25; First posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Ovarian Stimulation
MeSH Terms: interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMG group (Experimental): Induction of ovulation from 2nd day of cycle Follow diameter of follicle When follicle 18:22mm Receive HMG
  Interventions: Drug: HHMG
- H FSH plus HHMG (Experimental): Follow up ovulation from the 2nd day to 5th of menstruation cycle When follicle diameter 18mm to 22mm made induction of ovulation
  Interventions: Drug: HHMG

INTERVENTIONS:
Drug: HHMG — Induction of ovulation from the 2nd day of cycle to 5th day then follow the diameter of follicle Use transvaginal ultrasound When diameter of follicle 18 to 22 patients receiving HMG
  Other Names: Using HHMG for induction

SUMMARY:
Investigate and compare the efficacy of H FSH plus HMG Vs HMG alone on oocyte and embryo quality in IcsI patients

DETAILED DESCRIPTION:
70 patients divided in to 2groups Group A controlled ovarian stimulation with H FSH and HHMg Group B controlled ovarian stimulation with HMG alone Results will be discussed later

ELIGIBILITY:
Inclusion Criteria:

1. Infertil women aged from 20_35yr
2. Normal utreus
3. Normal ovaries
4. unexplained infertility
5. no endometriosis

Exclusion Criteria:

1 - poor responders to gonadotropin 2-Prior history of more than 3unsucceful ICSI 3-Any malformation of sexual organs

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 70 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Comparison between the efficacy of controlled ovarian stimulation with H FSH plus HMG Vs HmG alone on oocyte and embryo quality in IcsI patients | 9 months
  Comparison between the efficacy of controlled ovarian stimulation with H FSH plus HMG Vs HmG alone on oocyte and embryo quality in IcsI patients

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Ba Tarahony, Principal Investigator — Faculty of Medicine, Minia University